CLINICAL TRIAL: NCT03824938
Title: Aspirin for Exercise in Multiple Sclerosis (ASPIRE): A Double-Blind RCT of Aspirin or Acetaminophen Pretreatment to Improve Exercise Performance in Multiple Sclerosis (MS)
Brief Title: Aspirin for Exercise in Multiple Sclerosis (ASPIRE)
Acronym: ASPIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Victoria M. Leavitt, Assistant Professor, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AAAS2529; 1R21HD091836-01A1 (NIH)
Record Dates: First submitted 2019-01-09; First posted 2019-01-31 (Actual); Results first posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis
Keywords: exercise; aspirin; cooling; antipyretic
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Aspirin; Acetaminophen

STUDY DESIGN:
Intervention Model Description: This is a within-subject design double-blind RCT in which each participant receives 1 of 3 treatments at 3 timepoints (i.e., 3 separate days separated by 1-week washout periods).
Who Masked: Outcomes Assessor
Masking Description: Study biostatistician will derive the randomization schedule. Study pharmacy will make assignments and maintain blinding until data analysis is complete for the full sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Aspirin (Experimental): Aspirin 650 mg capsule by mouth, single dose
  Interventions: Drug: Aspirin 650mg Oral Capsule
- Acetaminophen (Active Comparator): Acetaminophen 650 mg capsule by mouth, single dose
  Interventions: Drug: Acetaminophen Tablet 650mg
- Placebo (Placebo Comparator): Placebo 650 mg capsule by mouth, single dose
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aspirin 650mg Oral Capsule — A 650mg dose of aspirin is administered in the laboratory one hour before participant completes a maximal exercise test.
  Other Names: Aspirin
  Arms: Aspirin
Drug: Acetaminophen Tablet 650mg — A 650mg dose of acetaminophen is administered in the laboratory one hour before participant completes a maximal exercise test.
  Other Names: Acetaminophen
  Arms: Acetaminophen
Other: Placebo — A placebo pill is administered in the laboratory one hour before participant completes a maximal exercise test.
  Arms: Placebo

SUMMARY:
This study investigates the use of aspirin as an exercise pre-treatment to reduce overheating and exhaustion, which may potentially allow many more people with multiple sclerosis to participate in and benefit from exercise. The design is double-blind, within-subject, with three arms: participants will receive one of three treatments at three separate study visits: aspirin, acetaminophen, and placebo, followed by completion of a maximal exercise test.

DETAILED DESCRIPTION:
Persons with multiple sclerosis benefit from exercise, but many avoid it because of exhaustion and overheating. This randomized controlled trial (RCT) tests aspirin as a method to increase time to exhaustion for persons with MS, through its antipyretic mechanism. Participants will be seen at our laboratory for maximal exercise tests on three separate days. At each session, they will be given one of three treatments: aspirin, acetaminophen (a drug that is anti-inflammatory but not antipyretic, thereby allowing for isolation of the antipyretic action of aspirin), and placebo. Primary outcome is increased time to exhaustion, secondary outcome is reduced body temperature increase during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing-remitting MS
* self-reported heat-sensitivity to exercise
* Expanded Disability Status Scale (EDSS) total score ≤ 6.0
* exacerbation-free (and no use of corticosteroids) for 6 weeks prior
* BMI ≤ 40

Exclusion Criteria:

* prior history of significant head injury, stroke, or other neurological disease/disorder
* current daily use of antipyretics or pain medication
* currently in a major depressive episode
* vascular disease of the legs, uncontrolled high blood pressure
* uncontrolled diabetes mellitus or problem with blood sugar levels
* contraindications to aspirin use (history of confirmed peptic ulcer, gastrointestinal or severe gynecological bleeding)
* tarry stool or known fecal occult blood
* uncontrolled syndrome of asthma, rhinitis, or nasal polyps
* contraindications to acetaminophen use (severe active hepatic disease, Hepatitis C Virus)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria M Leavitt, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw data for primary and secondary outcomes will be shared with qualified researchers upon reasonable request to study PI.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available from close of the study until 2031.
Access Criteria: Qualified researchers, upon request to study PI

REFERENCES:
- [Background] Leavitt VM, Blanchard AR, Guo CY, Gelernt E, Sumowski JF, Stein J. Aspirin is an effective pretreatment for exercise in multiple sclerosis: A double-blind randomized controlled pilot trial. Mult Scler. 2018 Oct;24(11):1511-1513. doi: 10.1177/1352458517739138. Epub 2017 Oct 27. PMID 29076760
- [Derived] Kever A, Nelson KE, Aguerre IM, Riley CS, Boehme A, Lee NW, Strauss Farber R, Levin SN, Stein J, Leavitt VM. ASPIRE trial: study protocol for a double-blind randomised controlled trial of aspirin for overheating during exercise in multiple sclerosis. BMJ Open. 2020 Nov 14;10(11):e039691. doi: 10.1136/bmjopen-2020-039691. PMID 33191260

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of the 97 screened, 60 were enrolled in the study.
Pre-assignment Details: Out of the 60 enrolled, 37 completed at least one visit.
Groups:
- Placebo First, Then Aspirin, Then Acetaminophen: First session: Placebo 650 mg capsule by mouth, single dose. A placebo pill is administered in the laboratory one hour before participant completes a maximal exercise test.
  Second session: Aspirin 650 mg capsule by mouth, single dose. A 650mg dose of aspirin is administered in the laboratory one hour before participant completes a maximal exercise test.
  Third session: Acetaminophen 650 mg capsule by mouth, single dose. A 650mg dose of acetaminophen is administered in the laboratory one hour before participant completes a maximal exercise test.
- Placebo First, Then Acetaminophen, Then Aspirin: First session: Placebo 650 mg capsule by mouth, single dose. A placebo pill is administered in the laboratory one hour before participant completes a maximal exercise test.
  Second session: Acetaminophen 650 mg capsule by mouth, single dose. A 650mg dose of acetaminophen is administered in the laboratory one hour before participant completes a maximal exercise test.
  Third session: Aspirin 650 mg capsule by mouth, single dose. A 650mg dose of aspirin is administered in the laboratory one hour before participant completes a maximal exercise test.
- Aspirin First, Then Placebo, Then Acetaminophen: First session: Aspirin 650 mg capsule by mouth, single dose. A 650mg dose of aspirin is administered in the laboratory one hour before participant completes a maximal exercise test.
  Second session: Placebo 650 mg capsule by mouth, single dose. A placebo pill is administered in the laboratory one hour before participant completes a maximal exercise test.
  Third session: Acetaminophen 650 mg capsule by mouth, single dose. A 650mg dose of acetaminophen is administered in the laboratory one hour before participant completes a maximal exercise test.
- Aspirin First, Then Acetaminophen, Then Placebo: First session: Aspirin 650 mg capsule by mouth, single dose. A 650mg dose of aspirin is administered in the laboratory one hour before participant completes a maximal exercise test.
  Second session: Acetaminophen 650 mg capsule by mouth, single dose. A 650mg dose of acetaminophen is administered in the laboratory one hour before participant completes a maximal exercise test.
  Third session: Placebo 650 mg capsule by mouth, single dose. A placebo pill is administered in the laboratory one hour before participant completes a maximal exercise test.
- Acetaminophen First, Then Placebo, Then Aspirin: First session: Acetaminophen 650 mg capsule by mouth, single dose. A 650mg dose of acetaminophen is administered in the laboratory one hour before participant completes a maximal exercise test.
  Second session: Placebo 650 mg capsule by mouth, single dose. A placebo pill is administered in the laboratory one hour before participant completes a maximal exercise test.
  Third session: Aspirin 650 mg capsule by mouth, single dose. A 650mg dose of aspirin is administered in the laboratory one hour before participant completes a maximal exercise test.
- Acetaminophen First, Then Aspirin, Then Placebo: First session: Acetaminophen 650 mg capsule by mouth, single dose. A 650mg dose of acetaminophen is administered in the laboratory one hour before participant completes a maximal exercise test.
  Second session: Aspirin 650 mg capsule by mouth, single dose. A 650mg dose of aspirin is administered in the laboratory one hour before participant completes a maximal exercise test.
  Third session: Placebo 650 mg capsule by mouth, single dose. A placebo pill is administered in the laboratory one hour before participant completes a maximal exercise test.
Period: Overall Study
Arm/Group | Placebo First, Then Aspirin, Then Acetaminophen | Placebo First, Then Acetaminophen, Then Aspirin | Aspirin First, Then Placebo, Then Acetaminophen | Aspirin First, Then Acetaminophen, Then Placebo | Acetaminophen First, Then Placebo, Then Aspirin | Acetaminophen First, Then Aspirin, Then Placebo
Started | 7 | 8 | 7 | 5 | 7 | 3
Completed | 5 | 6 | 7 | 3 | 6 | 2
Not Completed | 2 | 2 | 0 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: ASPIRE trial sample characteristics of the 37 active study participants.
Arm/Group | All Participants
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Time-to-exhaustion
Description: Duration of time exercising before reaching peak exertion, defined as cadence drop below 40 revolutions per minute (RPM) for >/= 5 seconds, or patient reaches volitional exhaustion in accordance with American Thoracic Society standard test termination criteria.
Time Frame: from start of exercise test until self-reported exhaustion, up to 30 minutes
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Placebo: Participants received placebo 650 mg capsule by mouth, single dose at any study visits, one hour before the initiation of the exercise test.
- Aspirin: Participants received aspirin 650 mg capsule by mouth, single dose at any study visits, one hour before the initiation of the exercise test.
- Acetaminophen: Participants received acetaminophen 650 mg capsule by mouth, single dose at any study visits, one hour before the initiation of the exercise test.
Arm/Group | Placebo | Aspirin | Acetaminophen
Number analyzed (Participants) | 32 | 31 | 32
seconds | 551.7 (78.4) | 331.6 (76.6) | 578.2 (82.1)

2. Primary Outcome: Exercise-induced Body Temperature Change
Description: Change in body temperature from pre- to post- maximal exercise test.
Time Frame: from start of exercise test until self-reported exhaustion, up to 30 minutes
Measure: Mean (Standard Deviation); unit: degrees Fahrenheit
Arm/Group | Placebo | Aspirin | Acetaminophen
Number analyzed (Participants) | 32 | 31 | 32
degrees Fahrenheit | 0.68 (0.35) | 0.006 (0.32) | 0.31 (0.35)

ADVERSE EVENTS:
Time Frame: Up to 30 days after study completion, an average of 4 weeks
Arm/Group | Placebo | Aspirin | Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT03824938/Prot_SAP_ICF_002.pdf